CLINICAL TRIAL: NCT06644963
Title: IMPELLA, Complications and Tolerance
Acronym: IMPACT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-08-120
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cardiogenic Shock
Keywords: Impella; pVAD; Bleeding; Thrombosis; hemocompatibily related adverse events
MeSH Terms: conditions — Shock, Cardiogenic; Hemorrhage; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Impella (5, 5.5 or CP) — Impella (5, 5.5 or CP) as an isolated circulatory support or combined with others Temporary Mechanical Circulatory Support

SUMMARY:
Myocardial infarction complicated by cardiogenic shock (AMICS) is associated with high morbidity and mortality, and devices like Impella® CP and Impella 5.0-5.5 are often used for hemodynamic support, either alone or combined with veno-arterial ECMO (ECMELLA). While recent studies suggest improved survival with Impella® in cardiogenic shock, complications remain common, particularly due to deep arterial access and the need for anticoagulation. Hemocompatibility-related adverse events (HRAEs) such as ischemia, bleeding (44%), hemolysis (32%), and stroke (13%) frequently occur. Achieving hemocompatibility between the patient's blood and the device is challenging, as pump flow, anticoagulation, and patient factors contribute to both thrombotic and hemorrhagic complications. Despite advances, further research is required to better understand and reduce these risks in clinical practice.

DETAILED DESCRIPTION:
Myocardial infarction complicated by cardiogenic shock (AMICS) is associated with high rates of morbidity and mortality. To provide hemodynamic support in these cases, intravascular microaxial left ventricular assist devices, such as Impella® CP and Impella 5.0-5.5, are frequently used, either alone in cardiogenic shock (CS) or in combination with veno-arterial ECMO (known as ECMELLA) for left ventricular unloading. Recent observational studies and randomized controlled trials have suggested improved survival rates with the use of Impella® in cardiogenic shock patients.

Despite the growing use of these devices, complications in clinical practice remain frequent. Due to the need for deep arterial access (14F for Impella CP and 21F for Impella 5.0) via femoral or axillary routes, as well as the necessity of anticoagulation, hemocompatibility-related adverse events (HRAEs) such as ischemic complications and bleeding are common, occurring in 18% and 44% of patients, respectively. Hemolysis has been reported in up to 32% of cases, while stroke affects up to 13%. Other less frequent complications include device deployment issues, pump thrombosis, implant site infections, and sepsis, all contributing to increased healthcare costs.

Achieving hemocompatibility between the patient's blood and the device remains a significant challenge despite advances in Impella technology. Balancing prothrombotic and prohemorrhagic forces at the blood/device interface is complex. This interface activates the coagulation cascade, generating a prothrombotic state, damaging von Willebrand multimers, and leading to hemolysis. The interplay of pump flow, pump speed, patient risk factors, and clinical management (anticoagulation) further complicates hemocompatibility, often resulting in thrombotic or bleeding events such as hemorrhagic stroke, circuit clots, or ischemic stroke.

Although the occurrence of HRAEs is well documented, particularly in the case of severe events like stroke, there is still an incomplete understanding of the factors driving these complications in modern clinical practice. Further research is needed to better delineate the risk factors and improve outcomes for patients receiving Impella support.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted for cardiogenic shock supported by Impella (5, 5.5 or CP) between January 1, 2010, and December 31, 2022 (as an isolated circulatory support or combined with others Temporary Mechanical Circulatory Support)

Exclusion Criteria:

* Absence of Impella
* Impella 2.5
* Impella RP (right)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted for cardiogenic shock supported by Impella (5, 5.5 or CP) between January 1, 2010, and December 31, 2022 (as an isolated circulatory support or combined with others Temporary Mechanical Circulatory Support)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Hemocompatibility related adverse events (HRAEs) | From start of hospitalization until hospital discharge, assessed up to 3 month
  Incidence of HRAEs with Impella (CP and/or 5 - 5.5) : Bleeding events (BARC >3b) and Thrombosis events ( ischemic stroke + pump thrombosis)

SECONDARY OUTCOMES:
Early mortality | From start of hospitalization until hospital discharge, assessed up to 3 month
  In-hospital all-cause mortality
Adverse events related to Impella devices | From start of hospitalization until hospital discharge assessed up to 3 month
  Hemolysis; Bacteremia; Infection of the device insertion site or the device itself
Duration of mechanical ventilation | From start of hospitalization until hospital discharge, assessed up to 3 month
  Total duration of invasive mechanical ventilation
Lengh of stay | From start of hospitalization until hospital discharge, assessed up to 3 month
  Total and in intensive care unit lenght of stay
Cardiac long-term project | From start of hospitalization until hospital discharge assessed up to 3 month
  Rate and % of patients with myocardial recovery, ventricular assist device or/and heart transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Aurore UGHETTO, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier university hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Van Edom CJ, Gramegna M, Baldetti L, Beneduce A, Castelein T, Dauwe D, Frederiks P, Giustino G, Jacquemin M, Janssens SP, Panoulas VF, Poss J, Rosenberg A, Schaubroeck HAI, Schrage B, Tavazzi G, Vanassche T, Vercaemst L, Vlasselaers D, Vranckx P, Belohlavek J, Gorog DA, Huber K, Mebazaa A, Meyns B, Pappalardo F, Scandroglio AM, Stone GW, Westermann D, Chieffo A, Price S, Vandenbriele C. Management of Bleeding and Hemolysis During Percutaneous Microaxial Flow Pump Support: A Practical Approach. JACC Cardiovasc Interv. 2023 Jul 24;16(14):1707-1720. doi: 10.1016/j.jcin.2023.05.043. PMID 37495347
- [Result] Vandenbriele C, Arachchillage DJ, Frederiks P, Giustino G, Gorog DA, Gramegna M, Janssens S, Meyns B, Polzin A, Scandroglio M, Schrage B, Stone GW, Tavazzi G, Vanassche T, Vranckx P, Westermann D, Price S, Chieffo A. Anticoagulation for Percutaneous Ventricular Assist Device-Supported Cardiogenic Shock: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 May 17;79(19):1949-1962. doi: 10.1016/j.jacc.2022.02.052. PMID 35550692
- [Result] Philipson DJ, Cohen DJ, Fonarow GC, Ziaeian B. Analysis of Adverse Events Related to Impella Usage (from the Manufacturer and User Facility Device Experience and National Inpatient Sample Databases). Am J Cardiol. 2021 Feb 1;140:91-94. doi: 10.1016/j.amjcard.2020.10.056. Epub 2020 Nov 2. PMID 33147430
- [Result] Amin AP, Spertus JA, Curtis JP, Desai N, Masoudi FA, Bach RG, McNeely C, Al-Badarin F, House JA, Kulkarni H, Rao SV. The Evolving Landscape of Impella Use in the United States Among Patients Undergoing Percutaneous Coronary Intervention With Mechanical Circulatory Support. Circulation. 2020 Jan 28;141(4):273-284. doi: 10.1161/CIRCULATIONAHA.119.044007. Epub 2019 Nov 17. PMID 31735078
- [Result] Dhruva SS, Ross JS, Mortazavi BJ, Hurley NC, Krumholz HM, Curtis JP, Berkowitz A, Masoudi FA, Messenger JC, Parzynski CS, Ngufor C, Girotra S, Amin AP, Shah ND, Desai NR. Association of Use of an Intravascular Microaxial Left Ventricular Assist Device vs Intra-aortic Balloon Pump With In-Hospital Mortality and Major Bleeding Among Patients With Acute Myocardial Infarction Complicated by Cardiogenic Shock. JAMA. 2020 Feb 25;323(8):734-745. doi: 10.1001/jama.2020.0254. PMID 32040163
- [Result] Moller JE, Engstrom T, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Frydland M, Holmvang L, Kjaergaard J, Sorensen R, Lonborg J, Lindholm MG, Udesen NLJ, Junker A, Schmidt H, Terkelsen CJ, Christensen S, Christiansen EH, Linke A, Woitek FJ, Westenfeld R, Mobius-Winkler S, Wachtell K, Ravn HB, Lassen JF, Boesgaard S, Gerke O, Hassager C; DanGer Shock Investigators. Microaxial Flow Pump or Standard Care in Infarct-Related Cardiogenic Shock. N Engl J Med. 2024 Apr 18;390(15):1382-1393. doi: 10.1056/NEJMoa2312572. Epub 2024 Apr 7. PMID 38587239